CLINICAL TRIAL: NCT06539897
Title: Effectiveness of Pelvic Floor Exercises and Sexual Education in Women Over 60: A Randomized Controlled Trial
Brief Title: Effectiveness of Pelvic Floor Exercises and Sexual Education in Women Over 60
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Alime Buyuk, PhD, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TBAEK-398
Record Dates: First submitted 2024-08-02; First posted 2024-08-06 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Sexual Dysfunction; Menopause; Pelvic Floor Disorders
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Pelvic Floor Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sexual Education Group (Experimental): The intervention group contains a combination of pelvic floor exercises and sexual education. One hour of each training consists of pelvic floor exercise practice and the other hour consists of sexual health education.
  Interventions: Behavioral: Sexual education
- No education (No Intervention): Women are not given information about sexual function

INTERVENTIONS:
Behavioral: Sexual education — These sessions of the sexual education program aim to increase women's knowledge and awareness about their own bodies. Women are informed about their own bodies, their identities, and the stages of sexual response, aiming to make the process clearer and more understandable. They will be encouraged to discover what sexuality means to them, their knowledge about sexuality will be questioned, and sexual myths, if any, will be revealed, and correct information about sexual myths will be provided to normalize sexuality. In addition, discussions will be held on the meanings of being a woman and an older woman, and women's perspectives on themselves and their self-esteem will be emphasized. In the third session, participants will be taught effective communication techniques to improve their communication skills with their partners.
  Arms: Sexual Education Group

SUMMARY:
Since the mid-19th century, "old age" has been increasingly recognized as a natural life stage, especially as the human lifespan extends. However, aging brings changes that negatively impact women's lives, causing diseases and lowering quality of life. Women now spend about one-third of their lives in old age. With 1.2 billion elderly women expected by 2030 (WHO), addressing aging issues is crucial for improving life quality. As life expectancy for women exceeds 80, advancements in modern and complementary medicine are making old age more bearable. Sexual health, closely tied to general health, should be considered in this context, involving both the woman and her family.

Aging leads to hormonal and muscle changes, causing pelvic floor dysfunctions such as incontinence, prolapse, constipation, and sexual dysfunction (Kikuchi, 2007). Pelvic floor muscles play a key role in sexual function, affecting lubrication, arousal, and orgasm (Berman et al., 2002; DeUgarte et al., 2004; Wright and O'Connor, 2015). Muscle tone imbalances can cause sexual pain disorders or decreased orgasm intensity and urinary incontinence (Berman et al., 2002; Berman, 2005; Mouritsen, 2009). Decreasing hormonal balance with age leads to issues like dyspareunia in women and erectile dysfunction in men (Kelley, 2018). Strategies like behavioral training and exercise can help mitigate age-related pelvic floor problems (Espunã-Pons, 2009).

DETAILED DESCRIPTION:
Since the mid-19th century, the concept of "old age" is frequently mentioned today, as the lifespan of humans, especially women, has been extended, and it is accepted as one of the natural and normal life stages of every woman. However, some changes that occur in old age negatively affect women's lives. This situation causes many diseases to emerge and decreases the quality of life of women (Yeni, 2004). Women will spend an average of one-third of their lives, and even longer in the future, in old age. According to the World Health Organization's estimate that 1.2 billion women will be elderly in 2030, knowing old age well and being able to overcome the problems it will create is the most important condition for increasing the quality of life of women over the age of 60. Today, when the average life expectancy for women is over 80, both the developments in the traditional approach of modern medicine and complementary medical developments have begun to make old age more bearable and allow for a dynamic life. Since Sexual Health is closely related to general health, it is most appropriate to approach sexuality in old age within the scope of old age, to plan the woman's life together with her and her family, and to take into account each parameter that will affect the quality of life (Taşkın, 2000). In parallel with the developments in the field of medicine, public health and the welfare of people in the last century, women's life expectancy has also increased. Today's women spend approximately 1/3 of their lives in the climacteric and post-climacterium period. In this respect, health problems related to this period are increasingly gaining great importance.

The decreasing and changing hormonal structure and muscle tissue changes with aging bring about pelvic floor dysfunctions. Especially factors such as the decrease in the volume of muscle tissue and its replacement by fat tissue and the decrease in the amount of estrogen/testosterone cause problems such as incontinence, prolapse, constipation and sexual dysfunctions (Kikuchi, 2007). Sexual dysfunction is also a frequently encountered condition in pelvic floor disorders in elderly individuals. Pelvic floor muscles, levator ani, bulbocavernosus and ischiocavernosus muscles, which are anatomical structures that have a direct effect on sexual function, regulate motor responses during vaginal penetration and orgasm, while the strength of these muscles increases lubrication, arousal and orgasm (Berman et al., 2002; DeUgarte et al., 2004; Wright and O'Connor, 2015). Excessive tone in these muscles causes sexual pain disorders; hypotonia seen in these muscles can lead to vaginal sensitivity, decreased orgasm intensity and urinary incontinence during sexual intercourse (Berman et al., 2002; Berman, 2005; Mouritsen, 2009). Especially with age, decreasing hormonal balance causes many problems such as dyspareunia in women and erectile dysfunction in men (Kelley, 2018). It has been reported that some strategies such as behavioral training, exercise or physical activity recommendations in pelvic floor dysfunctions minimize the problems that increase with age (Espunã-Pons M, 2009).

ELIGIBILITY:
Inclusion Criteria:

* Being in the age range of 60 and above
* Having good verbal communication skills
* Willing to participate in the study

Exclusion Criteria:

* Having severe musculoskeletal impairment
* Having a psychiatric disorder
* Having a neurogenic bladder
* Having malignancy in pelvic organs
* Having cognitive impairment

Ages: 60 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-08-02 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Pelvic Floor Impact Questionnaire (PFIQ-7) | 1 week
  Pelvic Floor Impact Questionnaire (PFIQ): The questionnaire has 7 questions and each question has 3 separate responses. The response to each item of satisfaction, impact and worry was rated from 3 (quite a bit) to 0 (not at all) for the PFIQ-7. The mean value for all the answered items within the corresponding scale (possible value 0-3) was estimated, then multiplied by (100/3) to obtain the scale score, range 0-100.
The Sexual Quality of Life-Female (SQOL-F) | 1 week
  The Sexual Quality of Life-Female (SQOL-F) questionnaire is a short instrument that specifically assesses the relationship between female sexual dysfunction and quality of life.
Pelvic Floor Distress Inventory PFDI-20 | 1 week
  Pelvic Floor Distress Inventory has a total of 20 questions and 3 scales (Urinary Distress Inventory, Pelvic Organ Prolapse Distress Inventory, and Colorectal-Anal Distress Inventory). Each short-form scale demonstrates significant correlation with their long-form scales
Arizona Sexuel Experiences Scale-ASEX | 1 week
  The ASEX scale is designed to measure five specific items identified in a comprehensive literature review as the core elements of sexual function: sexual drive, arousal, penile erection/vaginal lubrication, ability to reach orgasm, and satisfaction from orgasm.
The Sexual Self-Esteem Inventory for Women (SSEI-W) | 1 week
  The Sexual Esteem subscale is a part of the MSQ, and has been used widely in studies focusing on sexual esteem. The MSQ was developed by Snell et al. to measure psychological dimensions of sexuality, including 60 items and 12 subscales: sexual self-esteem, sexual preoccupation, internal sexual control, sexual consciousness, sexual motivation, sexual anxiety, sexual assertiveness, sexual depression, external sexual control, sexual monitoring, fear of sexual relations, and sexual satisfaction. These 12 dimensions are evaluated independently: they do not form a total score of sexual wellbeing based in all the 12 dimensions. Therefore, utilizing only one subscale such as sexual esteem, is not statistically problematic. The SEs consists of five items scaled from 0-4 (0=not at all, 1=slightly, 2=somewhat; 3=moderate, 4=very much). Higher scores correspond to greater mounts of the sexual esteem level

CONTACTS AND LOCATIONS:
Locations (1):
- Alime Buyuk, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Espuna-Pons M, Brugulat Guiteras P, Costa Sampere D, Medina Bustos A, Mompart Penina A. [Prevalence of urinary incontinence in Catalonia, Spain]. Med Clin (Barc). 2009 Nov 14;133(18):702-5. doi: 10.1016/j.medcli.2009.06.013. Epub 2009 Aug 5. Spanish. PMID 19656535
- [Background] Kikuchi A, Niu K, Ikeda Y, Hozawa A, Nakagawa H, Guo H, Ohmori-Matsuda K, Yang G, Farmawati A, Sami A, Arai Y, Tsuji I, Nagatomi R. Association between physical activity and urinary incontinence in a community-based elderly population aged 70 years and over. Eur Urol. 2007 Sep;52(3):868-74. doi: 10.1016/j.eururo.2007.03.041. Epub 2007 Mar 28. PMID 17412488
- [Background] Berman JR, Bassuk J. Physiology and pathophysiology of female sexual function and dysfunction. World J Urol. 2002 Jun;20(2):111-8. doi: 10.1007/s00345-002-0281-4. Epub 2002 Jun 1. PMID 12107542
- [Background] Wright JJ, O'Connor KM. Female sexual dysfunction. Med Clin North Am. 2015 May;99(3):607-28. doi: 10.1016/j.mcna.2015.01.011. Epub 2015 Mar 6. PMID 25841603
- [Background] Berman JR. Physiology of female sexual function and dysfunction. Int J Impot Res. 2005 Dec;17 Suppl 1:S44-51. doi: 10.1038/sj.ijir.3901428. PMID 16391543
- [Background] Mouritsen L. Pathophysiology of sexual dysfunction as related to pelvic floor disorders. Int Urogynecol J Pelvic Floor Dysfunct. 2009 May;20 Suppl 1:S19-25. doi: 10.1007/s00192-009-0831-z. PMID 19440779